CLINICAL TRIAL: NCT02950441
Title: Nicotinamide Adenine Dinucleotide and Skeletal Muscle Metabolic Phenotype (NADMet)
Brief Title: Nicotinamide Adenine Dinucleotide and Skeletal Muscle Metabolic Phenotype
Acronym: NADMet
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG_15-152
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2016-10

CONDITIONS: Aging
Keywords: Nicotinamide Riboside; Nicotinamide Adenine Dinucleotide; Skeletal muscle; Metabolism
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotinamide Riboside (Experimental): 1000mg (2x250mg tablets twice daily)
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Two tablets twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside
  Arms: Nicotinamide Riboside
Other: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to assess the physiological consequences of elevating Nicotinamide Adenine Dinucleotide (NAD+) availability using Nicotinamide Riboside (NR) supplementation in skeletal muscle tissue, and examine its effect upon muscle metabolic phenotype.

DETAILED DESCRIPTION:
-NAD+ sensitive metabolic decline in ageing, including sarcopenia, leads to a reduction in energy metabolism, contribute to chronic inflammation, disposing individuals to metabolic disease and overall decreased later-life health. Prominent metabolic changes include a decline in NAD+ content and deterioration in muscle NAD+ mediated signalling and mitochondrial function, ultimately compromising skeletal muscle and whole body energy homeostasis.

The most efficient means to boost NAD+ in muscle appears to be oral delivery of NR, and participants will be supplemented with 1000mg NR (2x x250mg tablets twice daily) for 3 weeks.

* Hypothesis: elevating skeletal muscle NAD+ bioavailability using NR supplementation will increase markers of mitochondrial function and that will manifest as a more favourable metabolic profile.
* Study Setting: the study will be carried out at the NIHR/Wellcome Trust Clinical Research Facility, Queen Elizabeth Hospital Birmingham.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 70-80 years
* BMI 20-30kg/m2
* Participants who are able to discontinue aspirin for 3 days prior to the muscle biopsy
* Participants who are able to discontinue statins and vitamin D supplements for a week before the second visit and for the duration of the study

Exclusion Criteria:

* Serious active medical conditions including inflammatory diseases or malignancies
* Significant past medical history including diabetes mellitus, ischaemic heart disease, cerebrovascular disease, significant respiratory disease requiring medication, epilepsy
* High blood pressure (BP>160/100mmHg)
* Oral Anticoagulants (like Warfarin, Dabigatran, Rivaroxaban) or Clopidogrel therapy which will increase the risk of bruising following a muscle biopsy

Ages: 70 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function assessment in skeletal muscle using high resolution respirometry | Following 3 weeks of NR supplementation
  Mitochondrial function assessment on muscle biopsies using high resolution respirometry
Skeletal muscle NAD+ levels in vastus lateralis biopsy using targeted metabolomics | Following 3 weeks of NR supplementation

SECONDARY OUTCOMES:
Improvement in response to oral glucose tolerance test/HOMA-IR | Following 3 weeks of NR supplementation
Improvement in lipid profile | Following 3 weeks of NR supplementation
Muscle Arterio-Venous Difference - Tissue-specific metabolite trafficking, oxygen consumption and CO2 production | Following 3 weeks of NR supplementation
Muscle biopsy: adaptive expression profile (genomic) | Following 3 weeks of NR supplementation
Changes in resting metabolic rate using indirect calorimetry | Following 3 weeks of NR supplementation
24 hour urine collection - NAD+ metabolomics and changes in steroid ratios using Gas chromatography/ mass spectrometry | Following 3 weeks of NR supplementation
Muscle strength - grip testing | Following 3 weeks of NR supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Lavery, PhD, Principal Investigator — Institute of Metabolism and Systems Research, University of Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No